CLINICAL TRIAL: NCT01500590
Title: Phase IV, Effect of Rennin-Angiotensin System Blockers on Glomerular Filtration Rate in Patients With Hypertension, Type 2 Diabetes With Normoalbuminuria--- A Randomized Controlled Trial
Brief Title: Effect of Renin-angiotensin System Blockers on Glomerular Filtration Rate in Patients With Hypertension, Type 2 Diabetes With Normoalbuminuria
Acronym: eGFR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2011-12-23; First posted 2011-12-28 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes; Hypertensive Disease
Keywords: Diabetes; hypertensive; without albuminuria
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Ramipril; Irbesartan; Amlodipine; Metoprolol; Indapamide; Methyldopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- renin-angiotensin system blockers (Experimental): Those eligible patients will be randomized into 2 groups. One group use renin-angiotensin systems (RAS) blockers to control their blood pressure, the other group will use other types of anti-hypertensive agents other than RAS blockers
  Interventions: Drug: Renin-angiotensin system blockers
- non-renin angiotensin system blockers (Active Comparator): These includes norvasc adalat retard natrilix betaloc aldomet
  amlodipine 2.5 to 10 mg once daily nifedipine retard 20mg once daily to 40mg twice daily indapamide 2.5mg once daily metoprolol 25mg to 100mg daily methyldopa 125 mg once daily to 500mg twice daily
  Interventions: Drug: non-renin angiotensin system blockers

INTERVENTIONS:
Drug: Renin-angiotensin system blockers — ramipril 2.5mg to 10mg once daily if patient experience cough, we will use irbesartan 150 mg to 300mg once daily
  Other Names: ramipril; irbesartan
  Arms: renin-angiotensin system blockers
Drug: non-renin angiotensin system blockers — amlodipine 2.5 to 10 mg once daily nifedipine retard 20mg to 40mg twice daily indapamide 2.5mg once daily metoprolol 25mg to 100mg daily methyldopa 125 mg to 500mg twice daily
  Other Names: norvasc, adalat retard, betaloc, natrilix or aldomet
  Arms: non-renin angiotensin system blockers

SUMMARY:
Diabetes is the leading cause of chronic kidney disease in developed countries. About 30-40% of patients with type 1 and type 2 diabetes mellitus will develop diabetic nephropathy. Microalbuminuria is often used as an early predictor of diabetic nephropathy. Many studies already demonstrated the renoprotective effect of Renin-angiotensin-system (RAS) blockers in patients with varying degree of albuminuria, few studies focus on studying the decline in glomerular filtration rate (GFR) among patients with normoalbuminuria. However a substantial number of diabetic patients exist with sub-normal GFR without microalbumin excretion. From literature, diabetes mellitus will have faster decline in GFR but the investigators do not know whether such decline can be slowed down by the use of RAS blockers as compared with other anti-hypertensive drugs. This Study investigate the effect of early treatment with RAS blockers on the decline rate of GFR in diabetic patients with normoalbuminuria.

DETAILED DESCRIPTION:
Renal excretory function, represented by GFR, deteriorates with age. After age 20-30 years, GFR declines by 1ml/min per year. This age related loss of renal function is proportional to blood pressure and glycemic level, and the rate of decline can accelerate up to 10-12 ml/min per year in poor BP and glycemia control.(1) Such rate of deterioration may lead to end-stage renal failure and the need for dialysis or transplantation.

Chronic kidney disease (CKD) is defined as either presence of kidney damage or GFR< 60 ml/min/1.73 m2 for more than 3 months. Kidney damage is defined as pathological abnormalities or markers of damage, including abnormalities in blood or urine tests or imaging studies. Microalbuminuria is often an early and sensitive marker of kidney damage in many types of chronic kidney disease. Among patients with chronic kidney disease, the stage is divided into stage 1-5 by the level of GFR, with higher stages representing lower GFR levels.(2) Renin-Angiotensin System ( RAS) is an enzymatic cascade in which angiotensinogen is cleaved by renin to form angiotensin I, which in turn, is converted by angiotensin converting enzyme (ACE) to form angiotensin II. Angiotensin II produces renal vasoconstriction, so blocking the RAS is shown to be a useful approach to reduce the renovascular risk. Among the RAS blocking agents, angiotensin converting enzyme inhibitor (ACEI) and angiotensin receptor blockers (ARB) are most commonly used in clinical practice.

Many studies already demonstrated the renoprotective effect of ACEI and ARB. These studies include MicroHOPE study(3), IRMA(4), IDNT(5), RENNAL(6) with subjects having varying degree of albuminuria. With compelling benefit of RAS blockers in diabetic patients with albuminuria, current guideline from American diabetic Association (ADA) recommend the use of ACEI and ARB to delay the progression of renal disease in diabetic nephropathy.(7) According to the National Kidney Foundation guideline, the workgroup recommend hypertensive patients with diabetes and CKD stage 1-4 should be treated with an ACEI or ARB, usually in combination with a diuretic.(8) For patients with suboptimal GFR (>= 60 ) without evidence of kidney damage like microalbuminuria, they are not considered as having CKD. There is lack of consensus on the selection of anti-hypertensive medication in this group of patients.

For subjects having normoalbuminuria, BENEDICT study demonstrates the delay in onset of microalbuminuria with the use of either trandolapril alone or trandolapril plus verapamil.(9) In ADVANCE trial, treatment with fixed combination of perindopril and indapamide reduced total renal event by 21%, defined as having new or worsening nephropathy or the development of new microalbuminuria.(10) However these studies mainly focus on using urinary albumin excretion as outcome measures. They seldom took the value of GFR into account.

However studies have found that significant decline in GFR in the absence of increase urine albumin excretion exists in a substantial percentage of adults with diabetes.(11) Decline in GFR should have diagnostic and prognostic value equivalent to urinary albumin excretion. However from literature, we cannot found the effect of RAS blockers on the decline in GFR. We therefore would like to carry out this study to investigate whether RAS blockers can delay the progress of renal disease, with particular attention to the value of GFR, in patients with GFR>=60 but without microalbuminuria.

ELIGIBILITY:
Inclusion criteria:

1. Age >=35 - 80 years old who is capable to give consent
2. Chinese
3. Either (i) Type 2 diabetes mellitus (DM) diagnosed according to ADA guideline or (ii) Hypertension defined as systolic blood pressure >140 or diastolic >90 mmHg or taking anti-hypertensive medication to attain blood pressure under these level or having (i) and (ii)
4. Estimated GFR (eGFR) (based on blood test taken 3 months prior to the date of consent) 60 - 89 ml/min/1.73m2 calculated by the abbreviated 4 variable Modification of Diet in Renal Disease (MDRD) study equation and no other identified causes of renal insufficiency.
5. Normoalbuminuria determined by urine albumin to creatinine ratio (based on urine test taken 3 months prior to the date of consent) <2.5 mg/mmol for men or <3.5 mg/mmol for women in first morning void urine sample.

Exclusion criteria:

1. Patients currently on ACEI or ARB as their anti-hypertensive medication
2. Pregnancy
3. Type 1 diabetes
4. Non-diabetic renal disease including renal artery stenosis
5. Secondary hypertension
6. History of symptomatic heart failure
7. History of myocardial infarction within 6 months
8. Specific indication for or contraindication to use ACEI or ARB
9. History of allergy to ACEI or ARB

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2011-11; Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
change of estimated GFR calculated by MDRD equation and onset of microalbuminuria | every 3 months
  Diabetes mellitus patients assigned to have RAS blockers have slower decline in GFR and delay in onset of microalbuminuria compared with those using other anti-hypertensive drugs. We measure the value of eGFR at baseline and every 6 months period in both control group and intervention group. The eGFR is calculated by MDRD equation. GFR = 186 x {serum creatinine (umol/l) /88.4}-1.154 x (age) -0.203 x ( 0.742 if female)
  We than calculate the difference of eGFR value every 6 month from the baseline. We would like to compare this difference in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Sing, Daniel CHU, M.B.,B.S., Principal Investigator — Hospital Authority, Hong Kong
Locations (1):
- Hospital Authority, HKEC, FM&PHC, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided